CLINICAL TRIAL: NCT02610907
Title: A Pilot Evaluation of Adhesives and How They Are Impacted by Out-put
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP265_01
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Ileostomy
MeSH Terms: interventions — Buffers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 01a (Experimental): This is a sub-study testing three patches consisting of an adhesive patch and a sleeve. The sleeve can contain one of three solutions:
  Buffer Own output Simulated output (digestive enzymes)
  All subjects will test the three solutions at the same time, hence the three patches with different solutions will be placed on the peristomal skin simultanously.
  Interventions: Other: Buffer; Other: Own output; Other: simulated output

INTERVENTIONS:
Other: Buffer — The sleeve contains phosphate buffered saline buffer
Other: Own output — The sleeve contains the subject own ileal effluent
Other: simulated output — The sleeve contains simulated output

SUMMARY:
The study investigates the impact real output (subjects own) and simulated output have on the adhesion of adhesives.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had an ileostomy for more than one year
4. Have intact skin on the area used in the evaluation
5. Has an ileostomy with a diameter up to (≤) 35 mm
6. Have a peristomal area accessible for application of patches/adhesive strips (assessed by investigating scientist)

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemotherapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Having dermatological problems in the peristomal- or abdominal area (assessed by investigating scientist)
5. Participating in other interventional clinical investigations or have previously participated in this evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Remaining adhesive area of adhesive | 30 hours
  The remaining adherent area of the adhesive is assessed by subtracting the area of output and swelling from the total adhesive area.

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Nielsen, MSc, Principal Investigator — R&D Principal Scientist
Locations (1):
- Coloplast A/S, Humlebæk, Denmark